CLINICAL TRIAL: NCT07248306
Title: Investigation of Temporomandibular Joint Function and Related Factors in Patients With Primary Sjögren's Syndrome
Brief Title: Temporomandibular Joint Dysfunction in Sjögren's Syndrome
Acronym: Sjögren
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Begüm AKAR, Principal investigator, Pamukkale University
Other Study IDs: Pamukkale U; Pamukkale University (Registry Identifier: Pamukkale University)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Sjogren Syndrome
Keywords: Sjogren syndrome; temporamandibular joint
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I: patients with primary Sjögren syndrome (pSS)
  Interventions: Diagnostic Test: Temporomandibular Joint Function

INTERVENTIONS:
Diagnostic Test: Temporomandibular Joint Function — Temporomandibular joint function and predictive parameters in patients with primary Sjögren Syndrome (pSS)

SUMMARY:
Study Purpose The purpose of this observational study is to determine the prevalence of temporomandibular dysfunction (TMD) in individuals diagnosed with Sjögren's syndrome and to examine the relationship between disease activity and TMD.

The main question to be answered is: Is TMD more common in individuals with Sjögren's syndrome, and is there a relationship between disease activity and TMD?

Method Participants diagnosed with Sjögren's syndrome will be evaluated. The prevalence and severity of TMD will be examined along with mouth opening, head posture, and oral health parameters.

ELIGIBILITY:
-Inclusion Criteria Individuals between 18 and 65 years of age. Must have a confirmed diagnosis of Sjögren's Syndrome. Must possess the mental capacity and education to understand the significance of the research.

Must be volunteers willing to participate in the study.

-Exclusion Criteria Incomplete questionnaires/scales. History of orthodontic treatment within the last six months. Presence of neurological or cognitive deficit. Patients with a history of pathology related to the temporomandibular joint (TMJ) and associated structures prior to the diagnosis of Sjögren's Syndrome.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Study Population: Women with Sjögren's Syndrome
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index (FAI) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Assesses the severity of TMD. As the score increases, the TMD severity (none, mild, moderate, severe) worsens. (0-15: None, 20-45: Mild, 50-65: Moderate, 70-100: Severe)
EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Evaluates disease activity. A high score (5 and above) indicates high disease activity. (The higher the average score, the more severe the symptoms of fatigue, pain, and dryness.)

SECONDARY OUTCOMES:
Xerostomia Inventory | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Measures the severity of dry mouth (xerostomia) symptoms. A higher score indicates more severe xerostomia symptoms.
Oral Health-Related Quality of Life - UK Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Assesses oral health-related quality of life. An increase in score generally indicates a greater deterioration in quality of life (i.e., worse oral health impact).
Visual Analog Scale (VAS) for Disease Involvement | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Numerically evaluates the severity of specific symptoms like dry mouth, dry eyes, facial skin dryness, and lip dryness. As the score approaches 10, the severity of dryness reaches its highest level.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Pamukkale, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No